CLINICAL TRIAL: NCT03160391
Title: Cognitive Effects of Music and Dance Training in Children: A Randomized Controlled Trial
Brief Title: Cognitive Effects of Music and Dance Training in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Melody Wiseheart, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: YorkU-MD1
Record Dates: First submitted 2017-05-06; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Cognitive Change

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Although the type of intervention provided was explicit (dance or music), participants, intervention providers, and outcomes assessors were not aware of the study hypotheses or predicted effects for each intervention. Hence they did not know whether they were in a treatment or control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Training (Experimental): Music Training
  Interventions: Behavioral: Music Training
- Dance Training (Active Comparator): Dance Training
  Interventions: Behavioral: Dance Training
- Passive control group (No Intervention): Passive control group

INTERVENTIONS:
Behavioral: Music Training — Training curriculums were developed using guidelines set by the Ontario Ministry of Education (The Ontario Curriculum, 2009) for teaching music to grades 1 to 3. Music was delineated into duration, pitch, dynamics and other expressive controls, timbre, texture/harmony, and form. training included direct instruction and group activities. All training programs had the same structure: a warm-up period, following by instruction from a teacher, and then group activities to practically demonstrate the concepts learned. Both programs involved working towards a variety of ensembles.
  Arms: Music Training
Behavioral: Dance Training — As with music training, dance was operationally defined by fundamental concepts for the art form, namely elements for body, space, time, energy, and relationship. The intervention involved both individual and group activities, with a combination of instruction and practical activities, and preparation for a final performance.
  Arms: Dance Training

SUMMARY:
The study used a randomized controlled trial to test the efficacy of two interventions (dance and musical training) for typically developing children. Interventions were run for three weeks in local community locations. Participants were tested before and after the intervention on a battery of cognitive and behavioural measures. They were compared across groups, and to a control group who do not receive the intervention.

The purpose of the current study was to assess the influence of dance and musical training on cognitive development. Research has indicated that musical training is associated with improve cognitive functioning, although the direction of such an association is unclear. Further, it is uncertain whether any benefits are specific to musical training or can also be demonstrated with other training activities. The current study used a randomized controlled trial to assess the causal effects of dance and musical training.

DETAILED DESCRIPTION:
Participants Monolingual children aged between six and nine years old were recruited from two local communities in Ontario, Canada. Children with developmental delays, learning disabilities, or previous arts training were excluded from the study.

Participants were randomly allocated to one of two groups

1. Dance intervention group
2. Music intervention group

To establish baseline performance levels and have a comparison, a passive control group was collected from the same towns using the same exclusion criteria.

Data analysis Difference scores were calculated for each measure by subtracting each participant's second testing session data from the first. When appropriate, iterative trimming with a 3 SD cutoff was used, by subject and by condition, to remove outliers. Results for each measure were analyzed using one-way ANOVAs (analysis of variance) for the between-subjects factor of training group (music, dance, or control).

ELIGIBILITY:
Inclusion Criteria:

* Monolingual

Exclusion Criteria:

* Developmental delays or learning disabilities
* Previous arts training (in dance, drama, or music)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Change in visuospatial working memory | Before and after intervention (3 weeks gap)
  Self-ordered pointing task (Cragg & Nation, 2007)
Change in interference control on flanker | Before and after intervention (3 weeks gap)
  Flanker task (Bunge, Dudukovic, Thomason, Vaidya, & Gabriela, 2002)
Change in color-shape task switching | Before and after intervention (3 weeks gap)
  color-shape task (Wiseheart, Viswanathan, & Bialystok, 2015)
Change in verbal working memory | Before and after intervention (3 weeks gap)
  Digit span (Weschler, 2008)
Change in interference control on Stroop | Before and after intervention (3 weeks gap)
  Stroop task (Cepeda, Blackwell, & Munakata, 2013)
Change in quantity-identity task switching | Before and after intervention (3 weeks gap)
  quantity-identity task (Cepeda, Cepeda, & Kramer, 2000)

SECONDARY OUTCOMES:
Change in processing speed using box completion | Before and after intervention (3 weeks gap)
  Box completion (Salthouse, 1993)
Change in Non-verbal intelligence | Before and after intervention (3 weeks gap)
  Kaufman Brief Intelligence Test (K-BIT-2; Kaufman & Kaufman, 2004)
Change in Receptive vocabulary | Before and after intervention (3 weeks gap)
  Peabody Picture Vocabulary Test (PPVT-IV; Dunn, Dunn, & Lenhard, 2015)
Change in processing speed using digit symbol | Before and after intervention (3 weeks gap)
  Digit symbol (Weschler, 1991)
Change in processing speed using symbol copy | Before and after intervention (3 weeks gap)
  Symbol copy (Weschler, 1991)

IPD SHARING:
Plan to Share IPD: Undecided